CLINICAL TRIAL: NCT03164629
Title: 3D Rotational CT Angiogram With Embolization Guidance and CBCT in Prostatic Artery Embolization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Siemens Corporation, Corporate Technology (Industry)
Responsible Party: Principal Investigator, Shivank Bhatia, Assistant Professor of Clinical Radiology & Urology, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20160589
Record Dates: First submitted 2017-05-22; First posted 2017-05-23 (Actual); Results first posted 2019-05-21 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Enlarged Prostate
Keywords: BPH; Lower Urinary Track Infection; Urine Retention
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- 3D Angiogram + Emboguide (Experimental): Participants will receive cone-beam CT 3D Emboguide: cone-beam CT with Embolization Guidance software (Emboguide) to identify prostatic arteries and assist endovascular navigation, by projecting a 3D road map of prostatic arteries on live fluoroscopy, in order to differentiate them from non-target vessels.
  Interventions: Device: cone-beam CT 3D Emboguide
- No 3D Angiogram + Emboguide (Active Comparator): Embolization will be guided by a standard of care CT.
  Interventions: Device: cone-beam CT 3D Emboguide

INTERVENTIONS:
Device: cone-beam CT 3D Emboguide — cone-beam CT with Embolization Guidance software (Emboguide) to identify prostatic arteries and assist endovascular navigation, by projecting a 3D road map of prostatic arteries on live fluoroscopy, in order to differentiate them from non-target vessels.

SUMMARY:
The purpose of this research study is to learn about how cone-beam Computerized Tomography scans (X-ray images taken from different angles) work together with an embolization guidance software (helps the doctor see the arteries that feed the prostate)to find and see arteries in the prostate.

ELIGIBILITY:
Inclusion Criteria:

* Patient is age 50 to 79, inclusive
* Patients undergoing Prostate artery embolization for BPH or urinary retention -Patient has signed informed consent.

Exclusion Criteria:

* Patients with biopsy proven prostate cancer
* Patient weight of >300 lbs

Ages: 50 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shivank Bhatia, Principal Investigator — University of Miami
Locations (1):
- Professional Arts Center, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 3D Angiogram + Emboguide: The following parameters will be recorded for the study group:
  Participants will receive cone-beam CT 3D Emboguide: cone-beam CT with Embolization Guidance software (Emboguide) to identify prostatic arteries and assist endovascular navigation, by projecting a 3D road map of prostatic arteries on live fluoroscopy, in order to differentiate them from non-target vessels.
Period: Overall Study
Arm/Group | 3D Angiogram + Emboguide | No 3D Angiogram + Emboguide
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3D Angiogram + Emboguide | No 3D Angiogram + Emboguide | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 12 | 26
  >=65 years | 11 | 13 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 25 | 25 | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Time for Prostatic Artery Catheterization
Description: For the cases using Emboguide this will be measured as the time from which the Emboguide is displayed on the live fluoroscopy to the time of prostatic artery catheterization. Emboguide display is in addition to the angiogram roadmap display.
  For the control cases this will be measured as the time from which the angiogram is displayed on the live fluoroscopy to the time of prostatic artery catheterization.
Time Frame: hour 2
Population: at times unable to catheterize the participants arteries
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | 3D Angiogram + Emboguide | No 3D Angiogram + Emboguide
Number analyzed (Participants) | 25 | 25
seconds
  Right Artery: number analyzed (Participants) | 25 | 24
  Right Artery | 273.40 (406.64) | 181.71 (185.11)
  Left Artery: number analyzed (Participants) | 24 | 24
  Left Artery | 206.38 (228.96) | 155.96 (216.32)

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- 3D Angiogram + Emboguide: articipants will receive cone-beam CT 3D Emboguide: cone-beam CT with Embolization Guidance software (Emboguide) to identify prostatic arteries and assist endovascular navigation, by projecting a 3D road map of prostatic arteries on live fluoroscopy, in order to differentiate them from non-target vessels.
Arm/Group | 3D Angiogram + Emboguide | No 3D Angiogram + Emboguide
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT03164629/Prot_SAP_000.pdf